CLINICAL TRIAL: NCT03726164
Title: A Study Investigating the Cardioprotective Benefits of Remote Ischaemic Postconditioning in Patients Presenting With Non ST Elevation Acute Coronary Syndromes Undergoing In-hospital Percutaneous Coronary Intervention
Brief Title: Remote Ischaemic Postconditioning in the Clinical Setting of NSTEACS and Urgent PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other); Surrey and Sussex Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/0138
Record Dates: First submitted 2017-05-08; First posted 2018-10-31 (Actual); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2017-05

CONDITIONS: Post Procedural Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote Conditioning group (Active Comparator): Patients will receive a standard remote ischaemia preconditioning protocol comprising a blood pressure cuff placed on arm and inflated to 200mmHg for 5 minutes and then deflated for 5 minutes, a cycle repeated three times, prior to the PCI procedure.
  Interventions: Device: Remote Conditioning
- Control Group (Placebo Comparator): Patients will receive a standard sham remote ischaemia preconditioning protocol with an un-inflated cuff be placed on the arm in this group of patients for 30 minutes. This is the sham intervention for this group.
  Interventions: Device: Sham protocol

INTERVENTIONS:
Device: Remote Conditioning — A Blood pressure cuff will be placed on the arm and inflated to 200mm hg for 5 minutes, and then deflated for 5 minutes, a cycle repeated 3 times.
  Other Names: RIC
  Arms: Remote Conditioning group
Device: Sham protocol — An un-inflated blood pressure cuff will be placed on the arm for 20 minutes.
  Other Names: Control
  Arms: Control Group

SUMMARY:
This study investigates the cardioprotective effect of remote ischaemic pre-/postconditioning in patients presenting with a NSTEMI/Unstable angina undergoing PCI.

DETAILED DESCRIPTION:
Patients presenting with Non ST elevation acute coronary syndromes (NSTEACS) - NSTEMI and Unstable angina patients are enrolled in this study.

Eligible patients are approached, with patient information sheets and are consented for involvement into the study. Patients are randomised to intervention or control. Patients randomised to intervention will receive 3 x 5 minutes of forearm ischaemia (with the cuff inflated to 200 mmHg) separated by 5 minutes of reperfusion between each cuff inflation, prior coronary angiography.

This protocol of episodic forearm ischaemia/reperfusion has been demonstrated to confer remote ischaemic preconditioning-induced protection.

Prior to the intervention, a blood sample will be taken to measure serum troponin T and CK-MB (baseline level). Following PCI patients will be reviewed on the wards and their ongoing recovery will be assessed and reviewed prior to discharge from the study. Troponin T and CK-MB levels will be measured for the 24 hours after PCI, at various time points (6 hour, 12 hour, 24 hour) as a measure of the degree of myocardial damage, and levels compared between the different treatment groups.

Primary end point

Myocardial injury (Peri-procedural Myocardial Infarction and Injury) measured by cTnT and CK-MB release over 24 hours after primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with NSTEMI/ Unstable angina undergoing percutaneous intervention

Exclusion Criteria:

* Known renal failure
* Known liver disease
* Peripheral vascular disease involving upper limbs
* Inability to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2008-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek M Yellon, PhD, FACC, Study Director — University College, London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remote Conditioning Group | Control Group
Started | 310 | 316
Completed | 99 | 119
Not Completed | 211 | 197

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Conditioning Group | Control Group | Total
Number analyzed (Participants) | 99 | 119 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.3) | 63.7 (11.0) | 62.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 30 | 44
  Male | 85 | 89 | 174
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 99 | 119 | 218

OUTCOME MEASURES:

1. Primary Outcome: Peri-Procedural Myocardial Injury
Description: Peri-Procedural Myocardial Injury will be assessed by the number of patients with peak troponin-T>3x 99th percentile upper reference limit
Time Frame: 24 hours post PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Remote Conditioning Group | Control Group
Number analyzed (Participants) | 99 | 119
Participants | 23 | 29

ADVERSE EVENTS:
Arm/Group | Remote Conditioning Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/119
Other Adverse Events (participants affected / at risk) | 0/99 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No